CLINICAL TRIAL: NCT05729997
Title: La música clásica en Directo y la Respuesta Frente a la Enfermedad y su evolución en Pacientes Con Insuficiencia Renal crónica
Brief Title: Live Classical Music and the Response to the Disease and Its Evolution in Patients With Chronic Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Miriam Serrano Soliva, mserranosoliva, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/0526
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Chronic Kidney Diseases; Haemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group listened for 4 weeks to live classical music during HD sessions lasting 30 to 40 minutes each.
  Interventions: Other: Listening to live classical music
- Control group (No Intervention): the control group carried out the usual treatment

INTERVENTIONS:
Other: Listening to live classical music — The group of musicians perform music in the hemodialysis room while patients receive treatment.
  Arms: Intervention group

SUMMARY:
People are most vulnerable to anxiety when faced with life-threatening situations such as illness, medical treatments and surgeries. When a person becomes ill, he and his family must face a series of changes in their life habits, must cope with admissions, aggressive treatments and endure physical pain. These changes can generate an unfavorable state of mind to face the disease, which sometimes worsens the previous clinical situation. The direct effect of music has been studied in different pathologies during the last years.

The proposed research sought to provide information on the influence of classical music listened to live and in situ in the hospital, and the response to the disease and its evolution, in patients with chronic renal failure. For this purpose, the effect of live music performances in hemodialysis rooms was analyzed and changes in the patients' mood and quality of life were observed. Changes in vital sign recording were also observed, all of which were assessed before and after the interventions. Finally, we checked if there were any changes in the variables described as confounders (KT/V-Albumin-Hemoglobin-Blood Pressure-Consumption of psychotropic drugs and analgesics), which could be attributable to listening to music.To test the effect in patients with chronic renal failure, live classical music was listened to in the hospital, as an adjuvant to treatment during haemodialysis processes. Ninety patients participated in 2 groups, the intervention group that listened to music during haemodialysis sessions and the control group that continued with their usual treatment. Changes in anxiety and mood were analyzed by means of the quality of life questionnaire (HAD) and quality of life by spheres with the KDQOL-SF questionnaire, before and after the intervention in both groups.

To test the effect in patients with chronic renal failure, live classical music was listened to in the hospital, as an adjuvant to treatment during haemodialysis processes. Ninety patients participated in 2 groups, the intervention group that listened to music during haemodialysis sessions and the control group that continued with their usual treatment. Changes in anxiety and mood were analyzed by means of the quality of life questionnaire (HAD) and quality of life by spheres with the KDQOL-SF questionnaire, before and after the intervention in both groups.

ELIGIBILITY:
Inclusion criteria:

* Patients over 18 years of age.
* Signed informed consent.
* To be more than 3 months in the chronic HD program.

Exclusion criteria:

* Inability to listen to music.
* Inability to answer the surveys.
* Failure to sign informed consent to participate.
* under 18 years of age.
* hospital admissions for more than 4 weeks or in the last two weeks of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Result variable:health-related quality of life (HRQL) | During the 1 month period, live musical performances were held in the HD rooms in two of the three weekly sessions. The musical sessions lasted about 30/40 min.
  Measured with the Kidney Diseasse health questionnaire Quality of life (KDQOL-SF) before and after the musical intervention.
  The scale includes 11 specific dimensions for kidney disease, the score for each dimension ranges from 0 to 100, where higher scores represent better health status, except in the specific scale of cognitive function and quality of social relationships where the highest score represents worse health status.
Result Variable: Anxiety and depression | During the 1 month period, live musical performances were held in the HD rooms in two of the three weekly sessions. The musical sessions lasted about 30/40 min.
  Measured whith the questionnaire Hospital Anxiety and Depression Scale (HAD) It is a self-administered questionnaire, composed of 14 questions divided into 2 subsections, one for the Anxiety scale (HAD-A) with 7 items and the other for the Depression scale (HAD-D) with 7 more items.
  For both scales, the score obtained results from the sum of each item, with the following ratings being considered in their evaluation
  * No case (NC) from 0 to 7
  * Doubtful Case (CD) from 8 to 10
  * Case (C) from 11 to the maximum value of 21.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital universitario y politecnica La Fe, Valencia, Spain

REFERENCES:
- [Result] Soliva, MS, Salvador, IR, Testal, AG, López, CC, Ramón, RO, Coca, JV, & Maset, RG (2022). Estudio de intervención para comprobar el efecto de la música clásica en directo durante la hemodiálisis sobre la calidad de vida de los pacientes con enfermedad renal crónica. nefrología , 42 (5), 559-567.
- See also: Related Info — https://doi.org/10.1016/j.nefro.2021.07.019